CLINICAL TRIAL: NCT07305935
Title: Comparative Efficacy of Early Caffeine Administration Versus Supportive Therapy in Preventing Acute Kidney Injury in Preterm Neonates
Brief Title: Comparison of Early Caffeine Administration Vs Supportive Therapy in Preventing Acute Kidney Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DR-NAZIA-MULTAN
Record Dates: First submitted 2025-12-05; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Caffeine; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Caffeine Group (Experimental): Neonates will receive caffeine citrate (IV or enteral) in 20 mg/kg loading dose within 24 hours of life, followed by a 5 mg/kg/day maintenance dose.
  Interventions: Drug: Caffeine
- Supportive Care Group (Experimental): Neonates will be given supportive care without caffeine
  Interventions: Drug: Supportive care

INTERVENTIONS:
Drug: Caffeine — Neonates will receive caffeine citrate (IV or enteral) in 20 mg/kg loading dose within 24 hours of life, followed by a 5 mg/kg/day maintenance dose.
  Arms: Early Caffeine Group
Drug: Supportive care — Neonates will be given supportive care without caffeine.
  Arms: Supportive Care Group

SUMMARY:
Recent observational data point towards a reduced incidence of acute kidney injury (AKI) with early caffeine use, but high-quality randomized controlled trials comparing early caffeine initiation to supportive therapy alone are lacking. This study aims to fill this critical gap by comparing the efficacy of early caffeine administration versus supportive therapy in preventing AKI in preterm neonates.

DETAILED DESCRIPTION:
There remains a debate about whether early initiation of caffeine therapy reduces the incidence and severity of AKI in preterm neonates compared to standard supportive care or not. Therefore, the incidence of AKI in preterm neonates will be compared between those receiving early caffeine therapy versus those receiving standard supportive therapy. The findings of this study would not only be a valuable addition to the statistics but also help clinicians to go for a better option in preterm neonates to prevent AKI, resulting in reducing the duration of mechanical ventilation, length of hospital stays, and all-cause neonatal mortality.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of any gender
* Neonates with gestational age <32 weeks
* Admitted within 6 hours of birth

Exclusion Criteria:

* Major congenital anomalies
* Severe birth asphyxia (Apgar <3 at 10 min)
* Pre-existing renal anomalies

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 14 days
  Incidence of AKI within the first 14 days of life.

SECONDARY OUTCOMES:
Duration of Acute Kidney Injury | Up to 30 days
  Time duration between onset of AKI and resolution.
Length of Hospital Stay | Up to 30 days
  Time duration from admission to discharge.
Mortality | Up to 30 days
  Mortality will be labelled when a patient expires during a hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Fatima, FCPS, Principal Investigator — The Children's Hospital & The Institute of Child Health, Multan; Rabia Saleem, FCPS, Principal Investigator — The Children's Hospital & The Institute of Child Health, Multan
Locations (1):
- The Children's Hospital & The Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.